CLINICAL TRIAL: NCT01248234
Title: Does Administration of Etomidate and Propofol if the Anesthetic Induction of the Elderly Hypertensive Patient Provide Superior Blood Pressure Stability in Response to Direct Laryngosacopy, When Compared to Propofol or Etomidate Alone?
Brief Title: Does Administration of Etomidate and Propofol of the Anesthetic Induction of Elderly Hypertensive Patient Provide Superior Blood Pressure Stability in Response to Direct Laryngoscopy When Compared to Propofol or Etomidate Alone?
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Did not begin
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2010-0097
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Hypertension
Keywords: elderly; hypertensive; anesthesia
MeSH Terms: conditions — Hypertension | interventions — Propofol; Etomidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Propofol (Active Comparator): Propofol alone will be used to put an elderly hypertensive patient to sleep for surgery.
  Interventions: Drug: propofol
- Etomidate (Active Comparator): Etomidate alone will be used to put an elderly hypertensive patient to sleep.
  Interventions: Drug: Etomidate
- Propofol and Etomidate (Active Comparator): A combination of Etomidate and Propofol will be used to put an elderly hypertensive patient to sleep for surgery.
  Interventions: Drug: Propofol and Etomidate

INTERVENTIONS:
Drug: propofol — Propofol 1mg/kg will be given once to put the patient to sleep for surgery.
  Arms: Propofol
Drug: Etomidate — Etomidate 0.3mg/kg will be given once to put the patient to sleep for surgery.
  Arms: Etomidate
Drug: Propofol and Etomidate — Etomidate 0.2mg/kg plus Propofol 0.5mg/kg will be given once to put the patient to sleep for surgery.
  Arms: Propofol and Etomidate

SUMMARY:
This study will attempt to show that a combination of drugs, Etomidate and Propofol, provide a more stable blood pressure when used to put elderly hypertensive patients to sleep than either drug used alone.

DETAILED DESCRIPTION:
Same as above.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 65 years old, with a history of hypertension.

Exclusion Criteria:

* Patients less than 65 years old or without a history of hypertension.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Blood pressure stability during anesthetic induction | 15 minutes
  Blood pressure will be measures every minute for 15 minutes following anesthetic induction

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Vaughn, MD, Study Chair — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States